CLINICAL TRIAL: NCT00393523
Title: A Study to Assess the Anamnestic Immune Response 4 to 8 Years After a Primary Vaccination Series With HBVAXPRO
Brief Title: Hepatitis B Vaccine Booster Study (V232-058)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V232-058; 2006_040
Record Dates: First submitted 2006-10-25; First posted 2006-10-27 (Estimated); Results first posted 2009-10-12 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- 5 µg Modified Process Hepatitis B Vaccine Booster (Group 1) (Active Comparator): Participants had previously received a primary series of 3 doses of RECOMBIVAX HB™ (5 µg (micrograms) per dose) during the first year of life outside of the context of the study.
  During this study, participants received a 5µg/0.5 ml dose of Modified Process Hepatitis B Vaccine (Booster Dose).
  Interventions: Biological: Comparator: Modified Process Hepatitis B Vaccine
- 10 µg ENGERIX-B™ Booster (Group 2) (Active Comparator): Participants had previously received a primary series of 3 doses of RECOMBIVAX HB™ (5 µg (micrograms) per dose) during the first year of life outside of the context of the study.
  During this study, participants received a dose of 10µg/per 0.5 ml ENGERIX-B™ (Booster Dose)
  Interventions: Biological: Comparator: Comparator: ENGERIX-B
- 5 µg Modified Process Hepatitis B Vaccine Booster (Group 3) (Active Comparator): Participants had previously received a primary series of 3 doses of ENGERIX-B™ (10 µg (micrograms) per dose) during the first year of life outside of the context of the study.
  During this study, participants received a 5µg/0.5 ml dose of Modified Process Hepatitis B Vaccine, (Booster Dose).
  Interventions: Biological: Comparator: Modified Process Hepatitis B Vaccine
- 10 µg ENGERIX-B™ Booster (Group 4) (Active Comparator): Participants had previously received a primary series of 3 doses of ENGERIX-B™ (10 µg (micrograms) per dose) during the first year of life outside of the context of the study.
  During this study, participants received a 10µg/0.5 ml dose of ENGERIX-B™ (Booster Dose).
  Interventions: Biological: Comparator: Comparator: ENGERIX-B
- 5 µg Modified Process Hepatitis B Vaccine (Group 5) (Experimental): Participants did not receive a prior vaccination with a hepatitis B vaccine.
  During the study, participants received a 5µg/0.5 ml dose of Modified Process Hepatitis B Vaccine.
  Interventions: Biological: Comparator: Modified Process Hepatitis B Vaccine

INTERVENTIONS:
Biological: Comparator: Modified Process Hepatitis B Vaccine — Single dose 5 µg/0.5ml modified process hepatitis B vaccine
  Arms: 5 µg Modified Process Hepatitis B Vaccine (Group 5); 5 µg Modified Process Hepatitis B Vaccine Booster (Group 1); 5 µg Modified Process Hepatitis B Vaccine Booster (Group 3)
Biological: Comparator: Comparator: ENGERIX-B — Single dose 10 µg/0.5ml ENGERIX-B
  Arms: 10 µg ENGERIX-B™ Booster (Group 2); 10 µg ENGERIX-B™ Booster (Group 4)

SUMMARY:
To assess the safety and immunogenicity of a booster dose of hepatitis B vaccine in children who have received a 3-dose primary series of either RECOMBIVAX HB or ENGERIX-B. The primary vaccination series (was given 4 to 8 years prior to study entry and consisted of a licensed hepatitis B vaccine product (either RECOMBIVAX HB or ENGERIX-B). The booster dose given in this study will be either an investigational Merck product (Modified Process Hepatitis B Vaccine) or licensed ENGERIX-B vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children 4 to 8 years of age
* Complete medical records documenting receiving a previous hepatitis B vaccination during the first year of life (for Cohort A and B only)
* Complete 3-dose vaccination with either a primary series of RECOMBIVAX HB or a primary series of ENGERIX-B (for Cohort A and B only)

Exclusion Criteria:

* Birth mother known to be a carrier of hepatitis B virus (Cohort C only)
* History of previous hepatitis B vaccine
* History of vaccination with any hepatitis B vaccine (Cohort C only)
* Known of suspected hypersensitivity to any component of RECOMBIVAX HB or ENGERIX-B (eg aluminum, yeast) recent administration of hepatitis B immune globulin (HBIg), serum immune globulin, or any other blood-derived product
* Receipt of investigational drugs or vaccines within 3 months prior to study vaccine or planned within study period
* Impairment of immunologic function or recent use of immunomodulatory medications
* A Combination of different hepatitis B vaccines used in the primary vaccination series (Cohort A and B only)

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1478 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Diez-Domingo J, Flores SA, Martin JC, Klopfer SO, Schodel FP, Bhuyan PK. A randomized, multicenter, open-label clinical trial to assess the anamnestic immune response 4 to 8 years after a primary hepatitis B vaccination series. Pediatr Infect Dis J. 2010 Oct;29(10):972-4. doi: 10.1097/INF.0b013e3181f1b3b6. PMID 20724955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 77 primary study sites in Spain and 1 study site in Canada.
  Date of first subject visit: 26-Sep-2006; Date of last subject visit: 23-June-2008
Pre-assignment Details: To be eligible for enrollment in the study, participants were to have received a primary series of 3 doses of the same type of hepatitis B vaccine (either RECOMBIVAX HB or ENGERIX-B) during the first year of life.
Groups:
- Modified Process Hepatitis B Vaccine Booster (Group 1): Participants received a primary series of 3 doses of RECOMBIVAX HB™ (5 µg (micrograms) per dose) during the first year of life outside of the context of the study; During the study, participants received one dose of Modified Process Hepatitis B Vaccine, 5 µg (micrograms) (Booster Dose)
- ENGERIX-B™ Booster (RECOMBIVAX-HB™ in Infancy) (Group 2): Participants received a primary series of 3 doses of RECOMBIVAX HB™ (5 µg (micrograms) per dose) during the first year of life outside of the context of the study; During the study, participants received one dose of ENGERIX-B™ (10 µg (micrograms) per dose) (Booster Dose)
- Modified Process Hepatitis B Vaccine Booster (Group 3): Participants received a primary series of 3 doses of ENGERIX-B™ (10 µg (micrograms) per dose).during the first year of life outside of the context of the study; During the study, participants received one dose of Modified Process Hepatitis B Vaccine, 5 µg (micrograms) (Booster Dose)
- ENGERIX-B™ Booster (ENGERIX-B™ in Infancy) (Group 4): Participants received a primary series of 3 doses of ENGERIX-B™ (10 µg (micrograms) per dose).during the first year of life outside of the context of the study; During the study, participants received one dose of ENGERIX-B™ (10 µg (micrograms) per dose) (Booster Dose)
- Modified Process Hepatitis B Vaccine (Group 5): Participants did not receive a prior vaccination with a hepatitis B vaccine; During the study, participants received one dose of Modified Process Hepatitis B Vaccine, 5 µg (micrograms)
Period: Overall Study
Arm/Group | Modified Process Hepatitis B Vaccine Booster (Group 1) | ENGERIX-B™ Booster (RECOMBIVAX-HB™ in Infancy) (Group 2) | Modified Process Hepatitis B Vaccine Booster (Group 3) | ENGERIX-B™ Booster (ENGERIX-B™ in Infancy) (Group 4) | Modified Process Hepatitis B Vaccine (Group 5)
Started | 376 | 375 | 353 | 354 | 20
Vaccination Visit 1 | 374 | 375 | 349 | 352 | 20
Completed | 364 | 366 | 349 | 348 | 19
Not Completed | 12 | 9 | 4 | 6 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1
Not completed — Protocol Violation | 6 | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 7 | 2 | 3 | 0
Not completed — Difficulties in specimen collection | 0 | 0 | 1 | 0 | 0
Not completed — Vaccine supply issue | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Process Hepatitis B Vaccine Booster (Group 1) | ENGERIX-B™ Booster (RECOMBIVAX-HB™ in Infancy) (Group 2) | Modified Process Hepatitis B Vaccine Booster (Group 3) | ENGERIX-B™ Booster (ENGERIX-B™ in Infancy) (Group 4) | Modified Process Hepatitis B Vaccine (Group 5) | Total
Number analyzed (Participants) | 376 | 375 | 353 | 354 | 20 | 1478
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.7 (0.92) | 5.7 (0.92) | 5.3 (1.05) | 5.4 (0.98) | 4.3 (0.66) | 5.5 (0.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 186 | 179 | 161 | 13 | 711
  Male | 204 | 189 | 174 | 193 | 7 | 767

OUTCOME MEASURES:

1. Primary Outcome: Antibody Response to Hepatitis B Surface Antigen in Subjects Who Received a 3-dose Primary Series of RECOMBIVAX HB in Infancy
Description: Number of subjects who received a 3-dose primary series of RECOMBIVAX HB™ in infancy and who demonstrated antibodies to hepatitis B surface antigen ≥10 mIU/mL at 4 weeks after receiving a booster dose of modified process hepatitis B vaccine or ENGERIX-B™.
Time Frame: 4 weeks after vaccination with either modified process hepatitis B vaccine or ENGERIX-B
Population: Per-protocol population (defined as the subjects that completed the study as defined by the protocol). Subjects were excluded from the analysis population mainly because they did not receive the primary series vaccination series as defined in the protocol or the study vaccine was not maintained at proper temperature as defined in the protocol.
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine Booster (Group 1) | ENGERIX-B™ Booster (RECOMBIVAX-HB™ in Infancy) (Group 2)
Number analyzed (Participants) | 340 | 333
Participants | 323 | 305
Statistical Analysis 1: Comparison: Modified Process Hepatitis B Vaccine Booster (Group 1); The primary purpose of this study was to show that subjects who received a primary series of RECOMBIVAX HB™ in the first year of life were adequately protected by RECOMBIVAX HB™ by measuring the immune response to a single booster dose of either a modified process vaccine or ENGERIX-B™; Test type: Superiority or Other; p < 0.001, Hochberg's step up — Adequate SPR required the lower bound of the 95.2% CI for the SPR for subjects in both Group 1 and Group 2 to be > 90% (P-Value < .024). Since only one group met the criteria, that group was retested at α=.012; The primary hypothesis was evaluated using Hochberg's step up approach to control multiplicity; Seroprotection rate (SPR) = 95.0, 95.2% CI [92.1 to 97.1] — Seroprotection rate (SPR)- defined as the percentage of subjects who demonstrate antibodies to hepatitis B surface antigen ≥10 mIU/mL
Statistical Analysis 2: Comparison: Modified Process Hepatitis B Vaccine Booster (Group 1); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Hochberg's step up — [p-value comment as in outcome 1, analysis 1]; The primary hypothesis was evaluated using Hochberg's step up approach to control multiplicity; Seroprotection rate (SPR) = 95.0, 97.6% CI [91.6 to 97.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: ENGERIX-B™ Booster (RECOMBIVAX-HB™ in Infancy) (Group 2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.19, Hochberg's step up — [p-value comment as in outcome 1, analysis 1]; The primary hypothesis was evaluated using Hochberg's step up approach to control multiplicity; Seroprotection rate (SPR) = 91.6, 95.2% CI [88.0 to 94.4] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Antibody Response to Hepatitis B Surface Antigen in Subjects Who Received a 3-dose Primary Series of ENGERIX-B in Infancy
Description: Number of subjects who received a 3-dose primary series of ENGERIX-B ™ in infancy and who demonstrated antibodies to hepatitis B surface antigen ≥10 mIU/mL at 4 weeks after receiving a booster dose of modified process hepatitis B vaccine or ENGERIX-B™.
Time Frame: 4 weeks after vaccination with either modified process hepatitis B vaccine or ENGERIX-B
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine Booster (Group 3) | ENGERIX-B™ Booster (ENGERIX-B™ in Infancy) (Group 4)
Number analyzed (Participants) | 338 | 328
Participants | 329 | 313
Statistical Analysis 1: Comparison: Modified Process Hepatitis B Vaccine Booster (Group 3); The purpose of the secondary analysis is to demonstrate that there is an adequate SPR in subjects who received a primary vaccination series of ENGERIX-B™ and a booster dose of modified process hepatitis B vaccine. An adequate response requires the lower bound of the two-sided 95% confidence interval for the SPR to exceed 90%; Test type: Superiority or Other; Seroprotection Rate (SPR) = 97.3, 95% CI [95.0 to 98.8] — Exact binomial confidence interval Seroprotection Rate (SPR)- defined as the percentage of subjects who demonstrate antibodies to hepatitis B surface antigen ≥10 mIU/mL

3. Other Pre Specified Outcome: Antibody Response to Hepatitis B Surface Antigen in Subjects Who Received a 3-dose Primary Series of RECOMBIVAX HB in Infancy
Description: Geometric Mean Titer (GMT) for all subjects who completed a 3-dose primary vaccination series of RECOMBIVAX HB™ and who received a booster dose of either modified process hepatitis B vaccine or ENGERIX-B™
Time Frame: 4 weeks after vaccination with either modified process hepatitis B vaccine or ENGERIX-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Modified Process Hepatitis B Vaccine Booster (Group 1) | ENGERIX-B™ Booster (RECOMBIVAX-HB™ in Infancy) (Group 2)
Number analyzed (Participants) | 340 | 333
mIU/mL | 476.9 [380.7 to 597.3] | 561.2 [435.6 to 723.1]

4. Other Pre Specified Outcome: Antibody Response to Hepatitis B Surface Antigen in Subjects Who Received a 3-dose Primary Series of ENGERIX-B in Infancy
Description: Geometric Mean Titer (GMT) for all subjects who completed a 3-dose primary vaccination series of ENGERIX-B™ and who received a booster dose of either modified process hepatitis B vaccine or ENGERIX-B™
Time Frame: 4 weeks after vaccination with either modified process hepatitis B vaccine or ENGERIX-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Modified Process Hepatitis B Vaccine Booster (Group 3) | ENGERIX-B™ Booster (ENGERIX-B™ in Infancy) (Group 4)
Number analyzed (Participants) | 338 | 328
mIU/mL | 1424.0 [1131.1 to 1792.8] | 1216.1 [923.6 to 1601.2]

ADVERSE EVENTS:
Description: Of the 1478 total participants in this study, 8 did not receive study vaccine, 17 received the incorrect study vaccine (different than what they were supposed to receive as part of the study), and 11 did not have safety follow-up information available. Thus, the total number of participants included in the safety analyses is 1442.
Arm/Group | Modified Process Hepatitis B Vaccine Booster (Group 1) | ENGERIX-B™ Booster (RECOMBIVAX-HB™ in Infancy) (Group 2) | Modified Process Hepatitis B Vaccine Booster (Group 3) | ENGERIX-B™ Booster (ENGERIX-B™ in Infancy) (Group 4) | Modified Process Hepatitis B Vaccine (Group 5)
Serious Adverse Events (participants affected / at risk) | 0/369 | 0/368 | 0/344 | 2/342 | 0/19
Other Adverse Events (participants affected / at risk) | 214/369 | 192/368 | 198/344 | 194/342 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modified Process Hepatitis B Vaccine Booster (Group 1) (N=369) | ENGERIX-B™ Booster (RECOMBIVAX-HB™ in Infancy) (Group 2) (N=368) | Modified Process Hepatitis B Vaccine Booster (Group 3) (N=344) | ENGERIX-B™ Booster (ENGERIX-B™ in Infancy) (Group 4) (N=342) | Modified Process Hepatitis B Vaccine (Group 5) (N=19)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modified Process Hepatitis B Vaccine Booster (Group 1) (N=369) | ENGERIX-B™ Booster (RECOMBIVAX-HB™ in Infancy) (Group 2) (N=368) | Modified Process Hepatitis B Vaccine Booster (Group 3) (N=344) | ENGERIX-B™ Booster (ENGERIX-B™ in Infancy) (Group 4) (N=342) | Modified Process Hepatitis B Vaccine (Group 5) (N=19)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 5 | 5 | 6 | 4 | 0
Motion Sickness (Ear and labyrinth disorders) | 1 | 0 | 1 | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 1 | 2 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 2 | 2 | 0
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye Swelling (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 9 | 4 | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 2 | 2 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 9 | 2 | 8 | 8 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 13 | 1 | 7 | 13 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Discomfort (General disorders) | 3 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 2 | 3 | 2 | 2 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 1 | 2 | 1 | 0
Pain (General disorders) | 1 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 22 | 20 | 17 | 32 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 3 | 2 | 3 | 6 | 0
Enterobiasis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 4 | 9 | 3 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 4 | 0 | 2 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 17 | 12 | 12 | 13 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Otitis media acute (Infections and infestations) | 2 | 0 | 3 | 1 | 0
Pharyngitis (Infections and infestations) | 11 | 4 | 5 | 4 | 0
Pharyngotonsillitis (Infections and infestations) | 2 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Scarlet fever (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 7 | 11 | 1 | 7 | 0
Tonsillitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 8 | 8 | 0
Varicella (Infections and infestations) | 0 | 1 | 2 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Bite (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0
Arthralgia (Metabolism and nutrition disorders) | 5 | 2 | 0 | 0 | 1
Bone pain (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Epiphysiolysis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0
Neck pain (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 0
Pain in extremity (Metabolism and nutrition disorders) | 5 | 0 | 3 | 0 | 0
Aphonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 16 | 18 | 19 | 14 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 10 | 22 | 12 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 9 | 5 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 4 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Bruising, Injection site for hepatitis B vaccine (General disorders) | 1 | 0 | 1 | 2 | 0
Erythema, Injection site for hepatitis B vaccine (General disorders) | 37 | 37 | 30 | 26 | 2
Hematoma, Injection site for hepatitis B vaccine (General disorders) | 0 | 3 | 3 | 3 | 0
Hypersensitivity, Injection site for hepatitis B vaccine (General disorders) | 0 | 2 | 3 | 2 | 0
Induration, Injection site for hepatitis B vaccine (General disorders) | 3 | 1 | 1 | 2 | 0
Edema, Injection site for hepatitis B vaccine (General disorders) | 1 | 0 | 0 | 0 | 0
Pain, Injection site for hepatitis B vaccine (General disorders) | 129 | 107 | 93 | 95 | 6
Paraesthesia, Injection site for hepatitis B vaccine (General disorders) | 0 | 0 | 1 | 1 | 0
Pruritus, Injection site for hepatitis B vaccine (General disorders) | 6 | 3 | 3 | 3 | 0
Scar, Injection site for hepatitis B vaccine (General disorders) | 0 | 0 | 1 | 0 | 0
Swelling, Injection site for hepatitis B vaccine (General disorders) | 54 | 38 | 40 | 25 | 3
Vesicles, Injection site for hepatitis B vaccine (General disorders) | 0 | 0 | 1 | 0 | 0
Warmth, Injection site for hepatitis B vaccine (General disorders) | 3 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.